CLINICAL TRIAL: NCT00578812
Title: A Prospective, Randomized, Controlled Clinical Investigation Comparing PCM® Cervical Disc Arthroplasty to Anterior Cervical Discectomy and Fusion: 2 Year Results From the US IDE Clinical Trial
Brief Title: PCM Cervical Disc System
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NuVasive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: G040081
Record Dates: First submitted 2007-12-19; First posted 2007-12-21 (Estimated); Results first posted 2013-02-12 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-06

CONDITIONS: Radiculopathy; Myelopathy
MeSH Terms: conditions — Radiculopathy; Spinal Cord Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PCM Cervical Disc - Investigational (Experimental): PCM Cervical Disc replacement at one level from C3 to T1
  Interventions: Device: PCM Cervical Disc
- ACDF - Control Group (Active Comparator): Anterior cervical discectomy and fusion (ACDF) at one level from C3 to T1
  Interventions: Device: Anterior Cervical Discectomy and Fusion (ACDF)

INTERVENTIONS:
Device: Anterior Cervical Discectomy and Fusion (ACDF) — Anterior cervical discectomy and fusion (ACDF) using a cervical plate and bone graft in patients with degenerated cervical discs and neurological symptoms at one level from C3 to T1
  Arms: ACDF - Control Group
Device: PCM Cervical Disc — PCM Cervical Disc replacement in patients with degenerated cervical discs and neurological symptoms at one level from C3 to T1
  Arms: PCM Cervical Disc - Investigational

SUMMARY:
The PCM Cervical Disc was studied in a prospective, multicenter, randomized FDA-approved investigational device exemption (IDE) clinical trial conducted in the United States to evaluate longitudinal outcomes over 2 years comparatively between the PCM Cervical Disc and anterior cervical discectomy and fusion (ACDF) with allograft and plate. Patients with adjacent or non-adjacent prior fusion were allowed. A total of 416 patients with a degenerated cervical disc at one level from C3-C4 to C7-T1 were enrolled in the clinical trial and 403 were treated. Patients were randomly assigned to be treated either with the PCM Cervical Disc or ACDF.

DETAILED DESCRIPTION:
The PCM Cervical Disc was studied in a prospective, multicenter, randomized FDA-approved investigational device exemption (IDE) clinical trial conducted in the United States to evaluate longitudinal outcomes over 2 years comparatively between the PCM Cervical Disc and anterior cervical discectomy and fusion (ACDF) with allograft and plate. Patients with adjacent or non-adjacent prior fusion were allowed. A total of 416 patients with a degenerated cervical disc at one level from C3-C4 to C7-T1 were enrolled in the clinical trial and 403 were treated. Patients were randomly assigned to be treated either with the PCM Cervical Disc or ACDF.

Patients were evaluated before surgery, during the operation, immediately after surgery, and then at 6 weeks, 3 months, 6 months, 12 months and 24 months, and yearly after surgery. The patients were recommended to have a physical therapy program for non-impact exercises and active range of motion exercises after surgery. Patients were also instructed to avoid repetitive cervical flexion and extension bending and lateral bending and rotation for 6 weeks following surgery.

The safety of the PCM Cervical Disc was assessed by comparing the adverse events, any additional surgical procedures, and the neurological outcomes to those in the ACDF control group. The effectiveness of the PCM Cervical Disc was assessed by evaluating patients' pain and function outcomes using a standard questionnaire, the Neck Disability Index (NDI), the severity of neck and arm pain based on a Visual Analog Scale (VAS) assessment, quality of life using a standard questionnaire, the Short Form-36 (SF-36), as well as a patient satisfaction questionnaire compared to the ACDF control group. In addition, the patients were evaluated using radiographic evaluations, including spinal range of motion, spinal disc height, device displacement or migration, spinal fusion status, and heterotopic ossification (abnormal bone formation).

The primary endpoint of the IDE trial was a composite measure termed "overall success," which was evaluated at 24 months postoperatively, and was defined as at least 20% improvement in neck disability index (NDI) from preoperative score; absence of reoperation, revision, or removal; maintenance or improvement in neurological status; and absence of radiographic or major complications during the 24-month follow-up period.

On October 26, 2012, the FDA granted Premarket Approval (PMA) for the PCM Cervical Disc. PCM Cervical Disc is indicated for use in skeletally mature patients for reconstruction of a degenerated cervical disc at one level from C3-C4 to C6-C7 following single-level discectomy for intractable radiculopathy (arm pain and/or a neurological deficit), with or without neck pain, or myelopathy due to a single-level abnormality localized to the disc space, and manifested by at least one of the following conditions confirmed by radiographic imaging (CT, MRI, X-rays): herniated nucleus pulposus, spondylosis (defined by the presence of osteophytes), and/or visible loss of disc height as compared to adjacent levels.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years;
* Diagnosis of radiculopathy or myelopathy of the cervical spine between C3-4 and C7-T1;
* Symptomatic at only one level from C3-C4 to C7-T1;
* Unresponsive to non-operative treatment for six weeks, or has the presence of progressive symptoms or signs of nerve root/spinal cord compression in the face of conservative treatment;
* Baseline NDI score of ≥30/100;
* Radiographically determined pathology at level to be treated correlating to primary symptoms, including at least one of the following: decreased disc height, degenerative spondylosis on CT or MRI, or disc herniation;
* Appropriate for treatment using an anterior surgical approach, including having no more than one previous anterior surgical approach to the cervical spine;
* Ability and willingness to comply with follow-up regimen; and
* Written informed consent given by subject or subject's legally authorized representative.

Exclusion Criteria:

* Infection at the site of surgery;
* History of, or anticipated treatment for, active systemic infection, including HIV infection or hepatitis C;
* Prior attempted or completed cervical spine surgery, except (1) laminoforaminotomy with less than one-third facetectomy at any level, or (2) a successful single-level anterior cervical fusion;
* More than one immobile vertebral level between C1-T1 from any cause, including but not limited to congenital abnormalities, osteoarthritic "spontaneous" fusions, and prior cervical spinal fusions;
* Previous trauma to the C3-T1 levels resulting in significant bony or disco-ligamentous cervical spine injury;
* Axial neck pain in the absence of other symptoms of radiculopathy or myelopathy justifying the need for surgical intervention;
* Radiographic confirmation of severe facet joint disease or degeneration.
* Osteoporosis:
* Severe diabetes mellitus requiring daily insulin management;
* Active malignancy: a history of any invasive malignancy (except non-melanoma skin cancer), unless the patient has been treated with curative intent and there have been no clinical signs or symptoms of the malignancy for at least 5 years;
* Tumor as source of symptoms;
* Symptomatic DDD or significant cervical spondylosis at two or more levels;
* Known or suspected allergy to cobalt, chromium, molybdenum, titanium, or polyethylene;
* Severe myelopathy to the extent that the patient is wheelchair bound;
* Pregnant (verified in patients of childbearing potential by a negative urine pregnancy test when preadmission testing is obtained), or interested in becoming pregnant during the duration of the study;
* Autoimmune disorders that impact the musculoskeletal system (e.g., lupus, rheumatoid arthritis; ankylosing spondylitis);
* Spinal axis disease (thoracic or lumbar) to the extent that surgical consideration is likely anticipated within 6 months after the cervical randomized procedure;
* Other degenerative joint disease (e.g. shoulder, hip, knee) to the extent that surgical consideration is likely anticipated within 6 months after the cervical randomized procedure;
* Previous spine surgery within the 6 months preceding the cervical randomized procedure;
* Current or recent history of substance abuse (drug or alcohol);
* Morbid obesity, defined as body mass index ("BMI") > 40 or more than 100 lbs. over ideal body weight;
* Currently using, or planning to use, bone growth stimulators in the cervical spine;
* Use of any other investigational drug or medical device within the last 30 days prior to surgery
* Currently a prisoner; or
* Currently pursuing personal litigation related to the neck or cervical spine injury; however, involvement in worker's compensation related litigation is not a required exclusion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 494 (Actual)
Dates: Start 2005-01; Primary Completion 2010-03 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (23):
- United States (23):
  - Tower Orthopedics, Beverly Hills, California
  - Spine Group Beverly Hills, Beverly Hills, California
  - Denver Spine, Greenwood Village, Colorado
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Midwest Orthopedic Associates at Rush, Chicago, Illinois
  - Chicago Back Institute, Chicago, Illinois
  - Goodman Campbell Brain and Spine, Indianapolis, Indiana
  - Towson Orthopedic Associates, Towson, Maryland
  - Wm. Beaumont Hospital, Southfield, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Columbia Orthopedic Research, Columbia, Missouri
  - Buffalo Spine Surgery, Lockport, New York
  - Institute for Spine Care, Syracuse, New York
  - The Cleveland Clinic, Cleveland, Ohio
  - OrthoNeuro, Westerville, Ohio
  - Neuroscience Specialists, Oklahoma City, Oklahoma
  - The Rothman Institute, Philadelphia, Pennsylvania
  - Neurosurgical Associates of San Antonio, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Virginia Brain and Spine, Winchester, Virginia
  - Olympia Othopaedic Associates, Olympia, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - NeuroSpine Center of Wisconsin, Appleton, Wisconsin

REFERENCES:
- See also: NuVasive — http://www.nuvasive.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Each clinical site could treat up to two (2) non-randomized investigational training patients prior to entering the randomized phase of the clinical trial.
Groups:
- PCM Cervical Disc - Investigational: PCM Cervical Disc replacement in patients with degenerated cervical discs and neurological symptoms at one level from C3 to T1
- Anterior Cervical Discectomy and Fusion - Control Group: Anterior cervical discectomy and fusion (ACDF) using a cervical plate and bone graft in patients with degenerated cervical discs and neurological symptoms at one level from C3 to T1
Period: Overall Study
Arm/Group | PCM Cervical Disc - Investigational | Anterior Cervical Discectomy and Fusion - Control Group
Started | 224 (Does not include investigational training patients (78 STARTED, 76 COMPLETED, 2 Not Treated).) | 192
Completed | 218 (Modified Intent-to-Treat (treated patients; analyzed as randomized).) | 185
Not Completed | 6 | 7
Not completed — Not treated | 6 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PCM Cervical Disc - Investigational | Anterior Cervical Discectomy and Fusion - Control Group | Total
Number analyzed (Participants) | 218 | 185 | 403
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.3 (9.0) | 43.7 (8.3) | 44.5 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 89 | 194
  Male | 113 | 96 | 209
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 202 | 170 | 372
  Black | 10 | 7 | 17
  Asian | 0 | 5 | 5
  Hispanic | 3 | 2 | 5
  Other | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 218 | 185 | 403

OUTCOME MEASURES:

1. Primary Outcome: Individual Patient Overall Success
Description: Individual patient overall success defined as ≥20% improvement in Neck Disability Index (NDI) from preoperative score, no device failures requiring revision, reoperation or removal, and the absence of radiographic or major complications during the 24-month follow-up period.
Time Frame: 24 Months
Population: Per Protocol
Measure: Number; unit: participants
Groups:
- PCM Cervical Disc-Investigational: PCM Cervical Disc replacement in patients with degenerated cervical discs and neurological symptoms at one level from C3 to T1
Arm/Group | PCM Cervical Disc-Investigational | Anterior Cervical Discectomy and Fusion - Control Group
Number analyzed (Participants) | 189 | 151
participants | 142 | 98

2. Secondary Outcome: Neck Pain Visual Analog Scale
Description: Improvement of ≥20mm in neck pain at 24 months compared to baseline.
Time Frame: 24 Months
Population: per protocol
Measure: Number; unit: participants
Arm/Group | PCM Cervical Disc - Investigational | Anterior Cervical Discectomy and Fusion - Control Group
Number analyzed (Participants) | 187 | 150
participants | 139 | 113

3. Secondary Outcome: Mean Neck Pain Visual Analog Scale
Description: Mean neck pain at 24 months on a 0-100 mm Visual Analog Scale (lower value is better).
Time Frame: 24 Months
Population: per protocol
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | PCM Cervical Disc - Investigational | Anterior Cervical Discectomy and Fusion - Control Group
Number analyzed (Participants) | 187 | 150
mm | 26.1 (28.7) | 30.4 (28.3)

4. Secondary Outcome: Worst Arm Pain Visual Analog Scale
Description: Improvement of ≥20mm in worst arm pain at 24 months compared to baseline.
Time Frame: 24 Months
Population: Per protocol
Measure: Number; unit: participants
Arm/Group | PCM Cervical Disc - Investigational | Anterior Cervical Discectomy and Fusion - Control Group
Number analyzed (Participants) | 187 | 150
participants | 148 | 113

5. Secondary Outcome: Mean Worst Arm Pain Visual Analog Scale
Description: Mean worst arm pain at 24 months on a 0-100mm Visual Analog Scale (lower value is better).
Time Frame: 24 Months
Population: Per protocol
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | PCM Cervical Disc - Investigational | Anterior Cervical Discectomy and Fusion - Control Group
Number analyzed (Participants) | 187 | 150
mm | 24.9 (29.2) | 27.5 (28.3)

6. Secondary Outcome: Clinically Significant Improvement on Neck Disability Index (NDI)
Description: Improvement in NDI of ≥20% at 24 months compared to baseline.
Time Frame: 24 Months
Population: Per protocol
Measure: Number; unit: participants
Arm/Group | PCM Cervical Disc - Investigational | Anterior Cervical Discectomy and Fusion - Control Group
Number analyzed (Participants) | 187 | 151
participants | 156 | 123

7. Secondary Outcome: Clinically Significant Improvement on Neck Disability Index (NDI)
Description: Improvement in NDI of ≥15-points at 24 months compared to baseline.
Time Frame: 24 Months
Population: Per protocol
Measure: Number; unit: participants
Arm/Group | PCM Cervical Disc-Investigational | Anterior Cervical Discectomy and Fusion - Control Group
Number analyzed (Participants) | 187 | 151
participants | 149 | 114

8. Secondary Outcome: Mean Neck Disability Index (NDI)
Description: Mean NDI at 24 months on a 0-100 scale (lower value is better).
Time Frame: 24 Months
Population: Per protocol
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PCM Cervical Disc - Investigational | Anterior Cervical Discectomy and Fusion - Control Group
Number analyzed (Participants) | 187 | 151
units on a scale | 21.8 (22.5) | 25.5 (21.5)

9. Secondary Outcome: Clinically Significant Improvement on SF-36 Physical Component Summary (PCS)
Description: Improvement of ≥15% on SF-36 PCS at 24 months compared to baseline.
Time Frame: 24 Months
Population: Per protocol
Measure: Number; unit: participants
Arm/Group | PCM Cervical Disc-Investigational | Anterior Cervical Discectomy and Fusion - Control Group
Number analyzed (Participants) | 187 | 151
participants | 133 | 98

10. Secondary Outcome: Mean SF-36 Physical Component Summary (PCS)
Description: Mean SF-36 PCS at 24 months on a 0-100 scale (lower value is better).
Time Frame: 24 Months
Population: Per protocol
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PCM Cervical Disc-Investigational | Anterior Cervical Discectomy and Fusion - Control Group
Number analyzed (Participants) | 187 | 151
units on a scale | 46.6 (11.0) | 45.0 (10.6)

11. Secondary Outcome: Clinically Significant Improvement on SF-36 Mental Component Summary (MCS)
Description: Improvement of ≥15% on the SF-36 MCS at 24 months compared to baseline.
Time Frame: 24 Months
Population: Per Protocol
Measure: Number; unit: participants
Arm/Group | PCM Cervical Disc-Investigational | Anterior Cervical Discectomy and Fusion - Control Group
Number analyzed (Participants) | 187 | 151
participants | 87 | 75

12. Secondary Outcome: Mean SF-36 Mental Component Summary (MCS)
Description: Mean SF-36 MCS at 24 months on a 0-100 scale (lower value is better).
Time Frame: 24 Months
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PCM Cervical Disc-Investigational | Anterior Cervical Discectomy and Fusion - Control Group
Number analyzed (Participants) | 187 | 151
units on a scale | 50.3 (11.1) | 49.3 (11.4)

13. Secondary Outcome: Dysphagia for Swallowing
Description: Mean dysphagia for swallowing at 24 months on a 0-100mm Visual Analog Scale (lower value is better).
Time Frame: 24 Months
Population: Per protocol
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | PCM Cervical Disc-Investigational | Anterior Cervical Discectomy and Fusion - Control Group
Number analyzed (Participants) | 183 | 147
mm | 8.8 (16.3) | 12.1 (20.1)

14. Secondary Outcome: Patient Satisfaction
Description: Mean Patient Satisfaction at 24 months on a 0-100 Visual Analog Scale (higher value is better).
Time Frame: 24 Months
Population: Per protocol
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | PCM Cervical Disc-Investigational | Anterior Cervical Discectomy and Fusion - Control Group
Number analyzed (Participants) | 182 | 146
mm | 82.8 (27.1) | 81.4 (25.7)

15. Secondary Outcome: Nurick's Classification of Disability (Myelopathy)
Description: Maintenance or improvement in Nurick's Classification from baseline to 24 months. Nurick's classification is a six-point scale, graded 0 to 5. A grade of 0 indicates no symptoms at all, while a grade of 5 is a bed or chair-bound patient. A patient "maintained" if their Nurick classification grade remained the same or "improved" if it decreased from baseline to 24 months.
Time Frame: 24 Months
Population: Per protocol with extended windows
Measure: Number; unit: participants
Arm/Group | PCM Cervical Disc-Investigational | Anterior Cervical Discectomy and Fusion - Control Group
Number analyzed (Participants) | 185 | 153
participants | 185 | 148

16. Secondary Outcome: Flexion/Extension Range of Motion at the Operative Level
Description: Mean flexion/extension range of motion at operative level at 24 months. The operative level is defined as the cervical spinal level at which the surgical procedure was performed.
Time Frame: 24 Months
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | PCM Cervical Disc-Investigational | Anterior Cervical Discectomy and Fusion - Control Group
Number analyzed (Participants) | 182 | 151
degrees | 5.7 (3.9) | 0.8 (0.8)

ADVERSE EVENTS:
Time Frame: Operative timepoint through 24 months.
Description: For AEs, Safety population used (all treated patients (pts) analyzed as-treated). One non-randomized investigational training pt and 4 randomized PCM pts were intraoperatively switched to receive ACDF so all included in ACDF group (N=190) and 4 randomized PCM pts were removed from randomized PCM group (N=214).
Arm/Group | PCM Cervical Disc-Investigational | Anterior Cervical Discectomy and Fusion - Control Group
Serious Adverse Events (participants affected / at risk) | 68/214 | 57/190
Other Adverse Events (participants affected / at risk) | 180/214 | 163/190
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PCM Cervical Disc-Investigational (N=214) | Anterior Cervical Discectomy and Fusion - Control Group (N=190)
Implant Related-Adjacent Level Disease (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4)
Implant Related - Implant Displacement/Loosening (Investigations) | 8 (8) | 0 (0)
Implant Related - Non Union (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Implant Related - Spinal Event (Injury, poisoning and procedural complications) | 3 (4) | 0 (0)
Implant Related - Subsidence (Investigations) | 1 (1) | 0 (0)
Implant Related - Trauma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Surgery Related - Neck/Arm Pain (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Surgery Related - Neurological (Nervous system disorders) | 2 (2) | 3 (3)
Surgery Related - Spinal Event (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Systemic - Cardiac Events (Cardiac disorders) | 3 (3) | 3 (3)
Systemic- Gastrointestinal (Gastrointestinal disorders) | 4 (5) | 2 (2)
Systemic - Infection (Infections and infestations) | 5 (5) | 3 (4)
Systemic - Mental Disorders (Psychiatric disorders) | 0 (0) | 3 (3)
Systemic - Musculoskeletal Trauma (Injury, poisoning and procedural complications) | 4 (4) | 8 (10)
Systemic - Musculoskeletal Adjacent Level Disease (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Systemic - Musculoskeletal / Back/Leg Pain (Musculoskeletal and connective tissue disorders) | 14 (18) | 5 (5)
Systemic - Musculoskeletal / Neck/Arm Pain (Musculoskeletal and connective tissue disorders) | 7 (10) | 8 (9)
Systemic - Musculoskeletal / Other (Musculoskeletal and connective tissue disorders) | 10 (10) | 2 (2)
Systemic - Musculoskeletal / Spinal Event (Musculoskeletal and connective tissue disorders) | 10 (10) | 11 (11)
Systemic - Neurologic (Nervous system disorders) | 0 (0) | 2 (2)
Systemic - Other (General disorders) | 7 (7) | 11 (11)
Systemic - Respiratory (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Systemic - Urogenital (General disorders) | 0 (0) | 6 (6)
OTHER ADVERSE EVENTS (reported when occurring in more than .5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PCM Cervical Disc-Investigational (N=214) | Anterior Cervical Discectomy and Fusion - Control Group (N=190)
Implant Related - Adjacent Level Disease (Musculoskeletal and connective tissue disorders) | 5 | 27
Implant Related - Non Union (Musculoskeletal and connective tissue disorders) | 0 | 11
Implant Related - Spinal Event (Musculoskeletal and connective tissue disorders) | 11 | 4
Surgery related - dysphagia/dysphonia (Injury, poisoning and procedural complications) | 14 | 23
Surgery related - Incision Site (Injury, poisoning and procedural complications) | 12 | 4
Surgery Related - Neck / Arm Pain (Injury, poisoning and procedural complications) | 21 | 32
Surgery Related - Neurologic (Nervous system disorders) | 12 | 10
Systemic - Gastrointestinal (Gastrointestinal disorders) | 12 | 6
Systemic - Infection (Infections and infestations) | 15 | 12
Systemic - Musculoskeletal Trauma (Injury, poisoning and procedural complications) | 42 | 32
Systemic - Musculoskeletal / Back/Leg Pain (Musculoskeletal and connective tissue disorders) | 36 | 33
Systemic - Musculoskeletal / Neck/Arm Pain (Musculoskeletal and connective tissue disorders) | 87 | 68
Systemic - Musculoskeletal / Other (Musculoskeletal and connective tissue disorders) | 29 | 17
Systemic - Musculoskeletal / Spinal Event (Musculoskeletal and connective tissue disorders) | 32 | 22
Systemic - Neurologic (Nervous system disorders) | 12 | 27
Systemic - Other (General disorders) | 42 | 26
Implant Related - Implant Displacement/Loosening (Investigations) | 10 | 1
Implant Related - Neck/Arm Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Implant Related - Other (General disorders) | 1 | 1
Implant Related - Radiolucency (Investigations) | 3 | 3
Implant Related - Subsidence (Investigations) | 1 | 2
Implant Related - Trauma (Injury, poisoning and procedural complications) | 1 | 1
Surgery Related - Gastrointestinal (Gastrointestinal disorders) | 2 | 2
Surgery Related - Infection (Infections and infestations) | 1 | 1
Surgery Related - Other (General disorders) | 4 | 7
Surgery Related - Respiratory (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Surgery Related - Spinal Event (Injury, poisoning and procedural complications) | 2 | 8
Surgery Related - Urogenital (General disorders) | 0 | 2
Surgery Related - Vertebral Fracture (Injury, poisoning and procedural complications) | 1 | 0
Systemic - Cardiac Events (Cardiac disorders) | 7 | 6
Systemic - Dysphagia/Dysphonia (General disorders) | 2 | 4
Systemic - Mental Disorder (General disorders) | 2 | 4
Systemic - Musculoskeletal/Adjacent Level Disease (Musculoskeletal and connective tissue disorders) | 2 | 1
Systemic - Other Trauma (Injury, poisoning and procedural complications) | 6 | 2
Systemic - Respiratory (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Systemic - Urogenital (General disorders) | 2 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators and Institutions will allow NuVasive to review and comment on any presentation or publication of any study information prior to its release to ensure such documents are accurate and do not disclose any trade secret or other confidential information. No information may be disclosed regarding the study without NuVasive's written permission.